CLINICAL TRIAL: NCT00417872
Title: Multicenter, Double Blind, Metronidazole Controlled, Dose Range Finding Study of Nitazoxanide in the Treatment of Clostridium Difficile Colitis
Brief Title: Study of Nitazoxanide in the Treatment of Clostridium Difficile Colitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Romark Laboratories L.C. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RM01-2015
Record Dates: First submitted 2007-01-03; First posted 2007-01-04 (Estimated); Last update posted 2007-01-04 (Estimated); Status verified 2005-10

CONDITIONS: Clostridium Difficile
Keywords: Clostridium difficile
MeSH Terms: interventions — nitazoxanide; Metronidazole

INTERVENTIONS:
Drug: Nitazoxanide
Drug: Metronidazole

SUMMARY:
The primary objective is to demonstrate non-inferiority of nitazoxanide administered 500 mg b.i.d compared to metronidazole administered 250 mg q.i.d. in resolving symptoms of Clotridium difficile colitis after seven days of treatment. Secondary objectives are to provide information on the times from first dose to last unformed stool and resolution of symptoms of colitis, the sustained response rates for the different tratment groups and the effect of treatment on Clostridium difficile toxin enzyme immunoassay/culture results during hospitalization.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years.
* In-patients with new onset of colitis evidenced by diarrhea (≥3 unformed stools within 24 hours), with one or more of the following: abdominal pain or cramps; peripheral leukocytosis, otherwise unexplained; or fever, otherwise unexplained.
* C. difficile toxin A or B detected in a stool specimen obtained within 7 days before enrollment by enzyme immunoassay.
* Patients able to take oral medications.
* Patients willing to avoid the following medications during the study: oral and intravenous metronidazole, oral vancomycin, anti-peristaltic drugs, opiates, Saccharomyces cerevisiae (baker's yeast), Lactobacillus GC, cholestyramine or colestipol. [Patients on opiates may be included in the study as long as they were taking opiates prior to enrollment and the dose is not increased during the study].
* Patients willing to abstain from alcohol during the 10-day treatment duration and for two days following treatment.

Exclusion Criteria:

* Patients with other known causes of diarrhea or colitis (e.g., Shigella, Salmonella, Cryptosporidium parvum, Giardia lamblia, Entamoeba histolytica, inflammatory bowel disease, irritable bowel syndrome, advanced AIDS or chemotherapy for malignancy).
* Use within 1 week of enrollment of any drug or therapy with anti-C. difficile activity such as oral or intravenous metronidazole and oral vancomycin. [Patients that have taken up to 2 doses of metronidazole or vancomycin can be included in the study].
* Females of child bearing age who are either pregnant, breast-feeding or not using birth control. A double barrier method, oral birth control pills administered for at least 2 monthly cycles prior to study drug administration, an IUD, or medroxyprogesterone acetate administered intramuscularly for a minimum of one month prior to study drug administration are acceptable methods of birth control for inclusion into the study. In addition, female patients of child-bearing potential should have a baseline pregnancy test and should agree to continue an acceptable method of birth control for the duration of the study (including follow-up).
* Patients taking phenytoin, celecoxib, and/or losartan. [Patients taking Coumadin® (warfarin) may be included as long the prothrombin time is monitored at least twice weekly during the first 2 weeks of the study and at least weekly thereafter].
* Patients with severe renal or hepatic impairment.
* Patients who are clinically unstable (e.g., patients with signs of toxic megacolon or imminent perforation).
* Serious systemic disorders incompatible with the study.
* History of hypersensitivity to metronidazole.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 114
Dates: Start 2004-01; Study Completion 2005-09

PRIMARY OUTCOMES:
Clinical response (resolution of all symptoms present at baseline) recorded on day 8

SECONDARY OUTCOMES:
Time from first dose to passage of last unformed stool
Time from first dose to resolution of symptoms
Sustained clinical response (resolution of all symptoms present at baseline with no recurrence during follow-up)
C. difficile toxin enzyme immunoassay/culture results during hospitalization

CONTACTS AND LOCATIONS:
Overall Officials: Ian M Baird, M.D., Principal Investigator — Remington-Davis Inc., and Riverside Infection Consultants, Inc.; Herbert L DuPont, M.D., Principal Investigator — CHI St. Luke's Health, Texas; Arvind K Gupta, M.D., Principal Investigator — Lehigh Valley Hospital; Robert S Jones, D.O., Principal Investigator — The Reading Hospital and Medical Center; Arnold L Lentnek, M.D., Principal Investigator — WellStar Infectious Diseases, Summit Surgical Specialists, and WellStar Kennestone Hospital; Daniel Musher, M.D., Principal Investigator — Houston Veterans Affairs Hospital; Fadi Saba, M.D., Principal Investigator — Bayfront Medical Center and Edward White Hospital
Locations (7):
- United States (7):
  - Bayfront Medical Center and Edward White Hospital, St. Petersburg, Florida
  - WellStar Infectious Diseases, Marietta, Georgia
  - Remington-Davis, Inc., and Riverside Infection Consultants, Inc., Columbus, Ohio
  - Lehigh Valley Hospital, Allentown, Pennsylvania
  - The Reading Hospital and Medical Center, West Reading, Pennsylvania
  - Houston Veterans Affairs Hospital, Houston, Texas
  - St. Luke's Episcopal Hospital, Houston, Texas